CLINICAL TRIAL: NCT01465607
Title: Implementation of an Efficacious Intervention for High Risk Women in Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas L. Patterson, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH087054 (NIH); R01MH087054 (NIH)
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: HIV; Syphilis; Gonorrhea; Chlamydia
Keywords: Condom use
MeSH Terms: conditions — Syphilis; Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theory-based counseling (Mujer Segura) (Experimental): Will consist of 40 FSWs at each of 12 clinics, randomized into this condition from a pool of 80 eligible participants.
  Interventions: Behavioral: Mujer Segura
- CENSIDA counseling program (didactic) (Active Comparator): Will consist of 40 FSWs at each of 12 clinics, randomized into this condition from a pool of 80 eligible participants.
  Interventions: Behavioral: CENSIDA counseling program

INTERVENTIONS:
Behavioral: Mujer Segura — Brief (35-minute) counseling intervention using techniques from Motivational Interviewing and principles of social cognitive theory (SCT) and theory of reasoned action (TRA).
  Arms: Theory-based counseling (Mujer Segura)
Behavioral: CENSIDA counseling program — Didactic HIV and STI counseling involving some personal risk assessment and presenting appropriate information on methods of transmission and for avoiding or reducing the risk of infection. Based on a counseling manual disseminated by CENSIDA, Mexico's federal HIV-AIDS prevention agency.
  Arms: CENSIDA counseling program (didactic)

SUMMARY:
This project seeks to determine the personal and organizational conditions that are most conducive to the widespread adoption by community-based organizations (CBOs) of effective programs for reducing the spread of HIV and other sexually transmitted infections (STIs). Taking a brief, single-session counseling program (called "Mujer Segura") that has been proven effective in reducing HIV and STIs in female sex workers who work in Mexican cities along the U.S. border, this project will study the implementation of the program in CBOs in 12 additional cities throughout Mexico to determine how best to ensure that the program remains true to the original model and retains its effectiveness. Mexico has been chosen because HIV is a global problem that respects no international borders, and because HIV prevention programs that can be implemented in settings with limited resources are urgently needed in many parts of the world.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Self-identify as female sex worker
* Exchanged sex for money, drugs, shelter, or other benefit in last 2 months
* Had unprotected anal or vaginal sex with male client at least once in last 2 months
* Agree to be tested for HIV & STIs at baseline and 6-month follow-u0

Exclusion Criteria:

* Previous positive HIV test result

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1228 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Reduction in HIV and STI incidence relative to control group | 6 months
  Female sex worker (FSW) participants will be tested at baseline and 6-month follow-up for HIV, syphilis, gonorrhea, and Chlamydia. Incidence rates for all infections at 6-month follow-up will be compared between the theory-based Mujer Segura group (N=40 per clinic) and the standard counseling group (N=40 per clinic).
Reduction in number of unprotected sex acts relative to control group | 6 months
  Female sex worker (FSW) participants will be assessed at baseline and 6-month follow-up using self-report measures of frequency of protected and unprotected sex acts with male clients. Changes in frequency at 6-month follow-up will be compared between the theory-based Mujer Segura group (N=40 per clinic) and the standard counseling group (N=40 per clinic).

SECONDARY OUTCOMES:
Fidelity to Mujer Segura intervention model | 6 months
  Counselors at each CBO will be assessed for their fidelity to the intervention protocol and assigned a numerical score. This number will be used to determine possible correlations between levels of fidelity and the efficacy of the Mujer Segura intervention at each clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Patterson, Ph.D., Principal Investigator — University of California, San Diego
Locations (4):
- Mexico (4):
  - Centro de Servicios Medicos (CSM) Revolucion, Mexico City, D.f.
  - CSM Guadalajara, Guadalajara, Jalisco
  - CSM Naranjos, Naranjos, Veracruz
  - CSM Veracruz, Veracruz, Veracruz

REFERENCES:
- [Derived] Pitpitan EV, Semple SJ, Aarons GA, Palinkas LA, Chavarin CV, Mendoza DV, Magis-Rodriguez C, Staines H, Patterson TL. Factors associated with program effectiveness in the implementation of a sexual risk reduction intervention for female sex workers across Mexico: Results from a randomized trial. PLoS One. 2018 Sep 11;13(9):e0201954. doi: 10.1371/journal.pone.0201954. eCollection 2018. PMID 30204761
- [Derived] Patterson TL, Semple SJ, Chavarin CV, Mendoza DV, Santos LE, Chaffin M, Palinkas LA, Strathdee SA, Aarons GA. Implementation of an efficacious intervention for high risk women in Mexico: protocol for a multi-site randomized trial with a parallel study of organizational factors. Implement Sci. 2012 Oct 29;7:105. doi: 10.1186/1748-5908-7-105. PMID 23107285